CLINICAL TRIAL: NCT04560686
Title: Phase II Study of Neoadjuvant Immune Checkpoint Blockade-Based Therapy With M7824 (Bintrafusp Alpha) for Untreated Resectable Non-Small Cell Lung Cancers
Brief Title: Bintrafusp Alfa Before Surgery for the Treatment of Untreated Resectable Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0910; NCI-2020-03769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0910 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-24; First posted 2020-09-23 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Resectable Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bintrafusp alfa, surgical resection) (Experimental): Patients receive bintrafusp alfa IV on days 1, 15, and 29 in the absence of unacceptable toxicity. Within 4-6 weeks after last dose of bintrafusp alfa, patients undergo surgery at the discretion of the treating surgeon. Within 8 weeks after surgery, patients may receive chemotherapy or undergo radiation therapy at the discretion of the treating physician.
  Interventions: Drug: Bintrafusp Alfa; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies how well bintrafusp alfa before surgery works in treating patients with non-small cell lung cancer for which the patient has not received treatment in the past (untreated) and that can be removed by surgery (resectable). Immunotherapy with bintrafusp alfa may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving bintrafusp alfa before surgery may help lower the risk of the cancer coming back after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the rate of major pathologic response (MPR).

OUTLINE:

Patients receive bintrafusp alfa intravenously (IV) on days 1, 15, and 29 in the absence of unacceptable toxicity. Within 4-6 weeks after last dose of bintrafusp alfa, patients undergo surgery at the discretion of the treating surgeon. Within 8 weeks after surgery, patients may receive chemotherapy or undergo radiation therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed previously untreated non-small cell lung cancer (NSCLC). If a diagnostic biopsy is available, a pre-treatment biopsy is not required. Patients with a suspected lung cancer are eligible, but pathology must be confirmed prior to initiating treatment on study. Neuroendocrine carcinomas (e.g. small cell lung cancer [SCLC], large cell neuroendocrine carcinoma, atypical carcinoid, carcinoid) are not eligible. Non-small cell carcinomas with neuroendocrine differentiation are eligible
* Patients with stage I-IIIA disease and IIIB (T3N2 only, and N2 single station), according to American Joint Committee on Cancer (AJCC) 8th edition, are eligible for arm A of the study. Patients with stage III, N2 single station, must not have more than one mediastinal lymph node station involved by tumor
* All patients must have lymph node evaluation of contralateral stations 2 and/or 4 to exclude N3 disease
* The patient must be a suitable candidate for surgery, in the opinion of the treating physician
* Predicted forced expiratory volume in 1 second (FEV1) >= 50%
* Predicted carbon monoxide diffusing capability test (DLCO) >= 50%
* Signed and dated written informed consent must be provided by the patient prior to admission to the study in accordance with International Conference on Harmonisation Good Clinical Practice (ICH-GCP) guidelines and to the local
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
* Absolute neutrophil count (ANC): >= 1.5 X 10^9 /L
* Hemoglobin: >= 9.0 g/dL
* Platelets >= 100 X 10^9 /L
* Total bilirubin: =< 1.5 X upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): =< 3 X ULN
* Creatinine: =< 1.5 X ULN or calculated creatinine clearance: >= 50 mL/min or 24-hour urine creatinine clearance: >= 50 mL/min

Exclusion Criteria:

* Mixed SCLC and NSCLC histology
* Major surgery within 4 weeks prior to the first dose of study intervention
* Thoracic radiation therapy (RT) of > 30 Gy within 6 months prior to the first dose of study intervention.
* Prior systemic therapy, including treatment with anti-PD-1/PD-L1 therapies and M7824, for treatment of the current lung cancer
* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug
* Previous malignant disease (other than the target malignancy to be investigated in this study) within the last 2 years. Participants with a history of cervical carcinoma in situ, superficial or noninvasive bladder cancer, or basal cell or squamous cell carcinoma in situ previously treated with curative intent are NOT excluded. Participants with other localized malignancies treated with curative intent need to be discussed with the principal investigator (PI) of the study
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant)
* Has interstitial lung disease (ILD) OR has had a history of pneumonitis that has required oral or IV steroids
* Pregnant or lactating female:

  * Women of childbearing potential (WOCB) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of immunotherapy.
  * Women of childbearing potential is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
* Unwillingness or inability to follow the procedures required in the protocol
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results. Participants with history of bleeding diathesis or recent major bleeding events considered by the Investigator as high risk for investigational drug treatment are also excluded
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* History of positive hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid indicating acute or chronic infection
* History of positive human immunodeficiency virus or known acquired immunodeficiency syndrome
* History of severe hypersensitivity reaction to any monoclonal antibody and/or to study drug components, any history of anaphylaxis, or recent (within 5 months) history of uncontrolled asthma
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Vaccine administration within 4 weeks of M7824 administration. Vaccination with live vaccines while on trial is prohibited. Administration of inactivated vaccines is allowed (for example, inactivated influenza vaccines)
* Patients who are sexually active, with preserved reproductive capacity, and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during and after the trial as detailed below:

  * WOCBP should use an adequate method to avoid pregnancy for 65 days after the last dose of investigational drug.
  * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.
  * Men receiving immunotherapy and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 125 days after the last dose of investigational product.
  * Women who are not of childbearing potential as well as azoospermic men do not require contraception
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cascone, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with stage I- IIIA NSCLC amenable for surgical resection were enrolled to this study in the Thoracic Medical Oncology Center at MD Anderson Cancer Center.
Pre-assignment Details: Two participants were consented; one screen failure. The trial was terminated earlier than planned due to an administrative decision taken by the PI/co-PI in collaboration with the study sponsor based on emerging data made available with the investigational agent being tested in other diseases in the perioperative setting.
Groups:
- Arm A: M7824 , Surgery, SOC Post-Op: M7824 1200 mg Q2 Weeks on D1, D15, & D29 followed by surgery, then possible SOC as post operative therapy
Period: Overall Study
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Major Pathologic Response (MPR)
Description: MPR will be defined as =< 10% viable tumor cells in the resected specimen using the methods described by Pataer et al. Will estimate the MPR rate with a 95% credible interval (CI) assuming that the MPR rate follows a prior beta distribution (0.5, 0.5) with one patient worth of information.
Time Frame: At time of surgery
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Adverse Events
Description: Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: Up to 1 year
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

3. Secondary Outcome: Peri-operative Morbidity and Mortality
Time Frame: Up to 1 year
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

4. Secondary Outcome: Response Rates to Induction
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 5 years post-treatment
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

5. Secondary Outcome: Recurrence-free Survival
Description: Will be computed using the Kaplan-Meier method.
Time Frame: At 12 months
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

6. Secondary Outcome: Recurrence-free Survival
Description: Will be computed using the Kaplan-Meier method.
Time Frame: At 18 months
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

7. Secondary Outcome: Recurrence-free Survival
Description: Will be computed using the Kaplan-Meier method.
Time Frame: At 24 months
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival
Description: Will be computed using the Kaplan-Meier method.
Time Frame: At 12 months
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

9. Secondary Outcome: Overall Survival
Description: Will be computed using the Kaplan-Meier method.
Time Frame: At 18 months
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Survival
Description: Will be computed using the Kaplan-Meier method.
Time Frame: At 24 months
Population: Data were not collected.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

11. Secondary Outcome: Complete Resection (RO) Rate
Description: Complete resection (R0) rate is defined as number of Participants that successfully underwent surgical resection with microscopically clear surgical margins.
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 1
Participants | 0

12. Secondary Outcome: Number of Participants With Pathologic Complete Response
Description: Pathologic complete response (pCR) in resected tumor specimens. pCR is defined as the absence of any viable residual tumor at the time of surgical resection in the primary lung lesion and lymph nodes, by central (core) pathology review.
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 1
Participants | 0

13. Secondary Outcome: CD8+ TILs in Resected Tumor Tissue
Description: Quantification of CD8+ TILs will be assessed by counting the cells positive for staining with an anti-CD8 antibody by immunohistochemistry and/or immunofluorescence in five random square areas (1 mm^2 each) in both intratumoral and peritumoral compartments using an automated system.
Time Frame: At time of surgery
Population: Due to Early termination of study no analysis was completed.
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Biomarker Analysis
Description: Multivariate analysis will be used to explore the role of biomarkers in predicting pathologic response to treatment, in an exploratory way.
Time Frame: Up to 5 years post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: from the time of the first protocol-specific intervention, until 100 days after the last dose of drug, unless the participant withdraws consent, approximately 11 months
Arm/Group | Arm A: M7824 , Surgery, SOC Post-Op
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: M7824 , Surgery, SOC Post-Op (N=1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: M7824 , Surgery, SOC Post-Op (N=1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Two participants were consented; one screen failure. The trial was terminated earlier than planned due to an administrative decision taken by the PI/co-PI in collaboration with the study sponsor based on emerging data made available with the investigational agent being tested in other diseases in the perioperative setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT04560686/Prot_SAP_000.pdf